CLINICAL TRIAL: NCT00021450
Title: Three Dimensional Conformal Radiotherapy / Intensity Modulated Radiotherapy Alone Vs Three Dimensional Conformal Therapy / Intensity Modulated Radiotherapy Plus Adjuvant Hormonal Therapy In Localized T1b-c, T2a, N0, M0 Prostatic Carcinoma. A Phase III Randomized Study
Brief Title: Radiation Therapy With or Without Bicalutamide and Goserelin in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-22991; EORTC-22991
Record Dates: First submitted 2001-07-13; First posted 2003-01-27 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Goserelin; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: bicalutamide
Drug: goserelin acetate
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Bicalutamide and goserelin may fight prostate cancer by reducing the production of testosterone. It is not yet known if radiation therapy is more effective with or without bicalutamide and goserelin in treating prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with or without bicalutamide and goserelin in treating patients who have localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the potential beneficial impact of radiotherapy with or without adjuvant bicalutamide and goserelin on the long-term outcome of patients with localized prostate cancer.
* Compare the acute and late radiation-induced side effects of these regimens in these patients.
* Compare the biochemical/clinical disease-free survival, overall survival, and time to local progression in patients treated with these regimens.
* Compare the time to clinical biological failure or death in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to tumor class (T1b-c vs T2a), initial prostate-specific antigen level (10 ng/mL vs 10-20 ng/mL vs greater than 20 ng/mL), Gleason score (2-6 vs 7-10) and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo 3-dimensional conformal radiotherapy or intensity-modulated radiotherapy once daily 5 days a week for 7-7.5 weeks.
* Arm II: Patients receive adjuvant oral bicalutamide once daily on days 1-30 and goserelin subcutaneously on days 8 and 98. Beginning on day 8, patients undergo radiotherapy as in arm I.

Quality of life is assessed at baseline and then at months 6, 12, 24, and 36.

Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 800 patients (400 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage II prostate cancer

  * T1b-c, N0, M0 with prostate-specific antigen (PSA) at least 10 ng/mL and/or Gleason score at least 7 (UICC 1997 classification) OR
  * T2a, N0, M0 (UICC 1997 classification)
* Serum PSA no greater than 50 ng/mL
* No involvement of pelvic lymph nodes

PATIENT CHARACTERISTICS:

Age:

* 80 and under

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other malignancy within the past 5 years except adequately treated basal cell skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No prior hormonal therapy

Radiotherapy:

* No prior pelvic radiotherapy

Surgery:

* No prior radical prostatectomy

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 819 (Actual)
Dates: Start 2001-04; Primary Completion 2008-04 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Biochemical and clinical disease-free survival as measured by Logrank prostate-specific antigen progression every 6 months until year 5, and annually thereafter

SECONDARY OUTCOMES:
Clinical disease-free survival as measured by Logrank every 6 months until year 5, and annually thereafter
Overall survival as measured by Logrank every 6 months until year 5, and annually thereafter
Local control as measured by Gray scale every 6 months until year 5, and annually thereafter
Acute toxicity as measured by NCI-CTC v2.0 up to 1 month post radiotherapy
Late toxicity as measured by EORTC and RTOG every 6 months until year 5, and annually thereafter
Quality of life as measured by EORTC QLQ-C30 and EORTC PR-25 every 6 months until year 5, and annually thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bolla, MD, Study Chair — CHU de Grenoble - Hopital de la Tronche
Locations (20):
- Belgium (3):
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - U.Z. Gasthuisberg, Leuven
- Bank Of Cyprus Oncology Centre, Nicosia, Cyprus
- Charles University Hospital, Hradec Králové, Czechia
- France (5):
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Centre Paul Strauss, Strasbourg
  - Centre d'Oncologie Saint-Yves, Vannes
- Saint Luke's Hospital, Dublin, Ireland
- Italy (2):
  - Spedali Civili di Brescia, Brescia
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
- Hopital de la Ville D'Esch-sur-Alzette, Esch-sur-Alzette, Luxembourg
- Netherlands (3):
  - Arnhems Radiotherapeutisch Instituut, Arnhem
  - University Medical Center Groningen, Groningen
  - Dr. Bernard Verbeeten Instituut, Tilburg
- Medical University of Gdansk, Gdansk, Poland
- Institut Catala d'Oncologia - Hospital Duran i Reynals, Barcelona, Spain
- Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland, United Kingdom

REFERENCES:
- [Background] Matzinger O, Poortmans P, Giraud JY, Maingon P, Budiharto T, van den Bergh AC, Davis JB, Musat E, Ataman F, Huyskens DP, Gulyban A, Bolla M; EORTC Radiation Oncology Group. Quality assurance in the 22991 EORTC ROG trial in localized prostate cancer: dummy run and individual case review. Radiother Oncol. 2009 Mar;90(3):285-90. doi: 10.1016/j.radonc.2008.10.022. Epub 2008 Nov 27. PMID 19038468
- [Result] Matzinger O, Duclos F, van den Bergh A, Carrie C, Villa S, Kitsios P, Poortmans P, Sundar S, van der Steen-Banasik EM, Gulyban A, Collette L, Bolla M; EORTC Radiation Oncology Group. Acute toxicity of curative radiotherapy for intermediate- and high-risk localised prostate cancer in the EORTC trial 22991. Eur J Cancer. 2009 Nov;45(16):2825-34. doi: 10.1016/j.ejca.2009.07.009. Epub 2009 Aug 12. PMID 19682889
- [Derived] Bolla M, Neven A, Maingon P, Carrie C, Boladeras A, Andreopoulos D, Engelen A, Sundar S, van der Steen-Banasik EM, Armstrong J, Peignaux-Casasnovas K, Boustani J, Herrera FG, Pieters BR, Slot A, Bahl A, Scrase CD, Azria D, Jansa J, O'Sullivan JM, Van Den Bergh ACM, Collette L; EORTC Radiation Oncology Group. Short Androgen Suppression and Radiation Dose Escalation in Prostate Cancer: 12-Year Results of EORTC Trial 22991 in Patients With Localized Intermediate-Risk Disease. J Clin Oncol. 2021 Sep 20;39(27):3022-3033. doi: 10.1200/JCO.21.00855. Epub 2021 Jul 26. PMID 34310202
- [Derived] Bolla M, Maingon P, Carrie C, Villa S, Kitsios P, Poortmans PM, Sundar S, van der Steen-Banasik EM, Armstrong J, Bosset JF, Herrera FG, Pieters B, Slot A, Bahl A, Ben-Yosef R, Boehmer D, Scrase C, Renard L, Shash E, Coens C, van den Bergh AC, Collette L. Short Androgen Suppression and Radiation Dose Escalation for Intermediate- and High-Risk Localized Prostate Cancer: Results of EORTC Trial 22991. J Clin Oncol. 2016 May 20;34(15):1748-56. doi: 10.1200/JCO.2015.64.8055. Epub 2016 Mar 14. PMID 26976418